CLINICAL TRIAL: NCT02936895
Title: The Effects of Vitamin D Supplementation in Respiratory Index of Severity in Children (RISC) of Hospitalized Patients With Community-acquired Pneumonia
Brief Title: Vitamin D Supplementation and Respiratory Index of Severity in Children (RISC) in Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Dr, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 188
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Low dose) (Experimental): vitamin D at a dose of 50,000 IU per day for 2 days
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Placebo (same size and shape) for 2 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — vitamin D at a dose of 50,000 IU per day for 2 days
  Other Names: cholecalciferol
  Arms: Vitamin D3 (Low dose)
Drug: Placebo — Placebo for 2 days
  Arms: Placebo

SUMMARY:
Childhood deaths from pneumonia is almost 2000 times higher in developing countries than in developed countries. In 1970, pneumonia was responsible for 9% of all deaths in children under 5 years. This rate was 2% in 2007.

Some studies have shown that supplementing with vitamin D reduces disease of the respiratory tract infection. Some other studies have shown anti-inflammatory effect of vitamin D in cell lines. Studies about the role of vitamin D supplementation in pneumonia in children are inadequate to conclude about its role.

The aim of this study is to determine the efficacy of vitamin D supplementation in Respiratory Index of Severity in Children (RISC) hospitalized clinical outcomes of hospitalized patients with community-acquired pneumonia.

ELIGIBILITY:
Inclusion criteria

* Aged between 2 months to 6 years
* Definite diagnosis of pneumonia

Exclusion criteria

* Immunocompromised patients
* Airway hypersensitivity or asthma
* allergies
* nasal polyps
* Using inhaled medications to one month prior to the study
* Receiving high doses of vitamin D
* Avoiding to complete informed consent form

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Respiratory Index of Severity in Children (RISC) | through study completion, an average of 4 days
  For determining severity of pneumonia, RISC (Respiratory Index of Severity in Children) scoring system was used, including oxygen saturation, chest retraction, wheezing and refusal to feed, and also contains standards growth (weight for age).

SECONDARY OUTCOMES:
Duration of hospitalization | through study completion, an average of 4 days
  Duration of hospitalization of the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Mohammadi hospital, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: No